CLINICAL TRIAL: NCT05086406
Title: Virtual and Video Counseling Versus In-Office Counseling for Laparoscopic Hysterectomy: A Randomized Controlled Trial
Brief Title: Virtual and Video Counseling Versus In-Office Counseling for Laparoscopic Hysterectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FLA 21-022
Record Dates: First submitted 2021-10-01; First posted 2021-10-20 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Patient Engagement
Keywords: Patient Preparedness; Total Laparoscopic Hysterectomy; Pre-operative Education; Virtual Visits/Counseling
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Intervention Model Description: Patients undergoing a laparoscopic hysterectomy for benign gynecologic etiologies with Drs. Arnolds, Frazzini Padilla, or Sprague at Cleveland Clinic Florida Section of Minimally Invasive Gynecologic Surgery will be recruited at the visit where decision is made to proceed with surgery. Enrolled subjects will be randomized using a computer generator into either the control group or the study group. Subjects will be notified of which group they have been selected to at the time of scheduling for their pre-operative visit. The control group will undergo standard in-office pre-operative counseling visit. The study group will receive pre-operative counseling via video followed by a virtual visit with a gynecologic surgery provider, using standard and secure communications that are currently approved by Cleveland Clinic. The link to the video and instructions for the virtual visit will be sent to the subject either via email and/or through a message on the electronic medical record platform.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-Office Visit Group (No Intervention): This control group will undergo standard in-office pre-operative counseling visit.
- Virtual Visit Group (Experimental): This study group will receive pre-operative counseling via video, created by the Department of Gynecology at Cleveland Clinic Florida, followed by a virtual visit with a gynecologic surgery provider.
  Interventions: Other: Combination of Video and Virtual Pre-operative Counseling

INTERVENTIONS:
Other: Combination of Video and Virtual Pre-operative Counseling — Intervention will be a pre-operative counseling video followed by a virtual visit with a gynecologic surgery provider, using standard and secure communications.
  Arms: Virtual Visit Group

SUMMARY:
Compare preparedness for total laparoscopic hysterectomies between patients who undergo virtual visits and those who undergo in-office visits for pre-operative counseling.

DETAILED DESCRIPTION:
The proposed research study looks to evaluate the effectiveness of combination of video counseling and virtual visits for pre-operative counseling as compared to in-office pre-operative counseling visits ahead of total laparoscopic hysterectomy surgery. Comparison of the two cohorts will be based on responses to surveys regarding patient preparedness on the day of surgery and information obtained from the electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing laparoscopic hysterectomy for benign gynecologic etiologies.
* Age of 20 years or older
* Understand English language (written and spoken) without difficulty

Exclusion Criteria:

* Age less than 20 years old
* Diagnosis of malignancy
* No access to technology that would allow for watching counseling video and/or completion of virtual visit

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Differences in patient preparedness | Up to time of surgery
  Assess differences in patient preparedness at the time of the surgery between patients who received video and virtual pre-operative counseling versus those who received in-person counseling.

SECONDARY OUTCOMES:
Unplanned office or emergency department visit | Up to 6 weeks after surgery
  Observe how many patients from each cohort require an unplanned visit to the office or visit to the emergency department.
Same-day discharge versus admission rates | Up to 1 day after surgery
  Note differences in same-day discharges or admission rates following surgery between each cohort
Readmission rates | Up to 6 weeks after surgery
  Record differences in readmission rates in the 6 week post-operative period between each cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Arnolds, MD, Principal Investigator — Cleveland Clinic Florida Gynecology
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers. The goal of the study is to look at outcomes of each cohort and it is not necessary to analyze each IPD.

REFERENCES:
- [Background] Krantz TE, Rogers RG, Petersen TR, Dunivan GC, White AB, Madsen AM, Jeppson PC, Ninivaggio CS, Cichowski SB, Komesu YM. Peer-Centered Versus Standard Physician-Centered Video Counseling for Midurethral Sling Surgery: A Randomized Controlled Trial. Female Pelvic Med Reconstr Surg. 2020 Aug;26(8):470-476. doi: 10.1097/SPV.0000000000000784. PMID 31596774
- [Background] Greene KA, Wyman AM, Scott LA, Hart S, Hoyte L, Bassaly R. Evaluation of patient preparedness for surgery: a randomized controlled trial. Am J Obstet Gynecol. 2017 Aug;217(2):179.e1-179.e7. doi: 10.1016/j.ajog.2017.04.017. Epub 2017 Apr 18. PMID 28431952
- [Background] Fountain CR, Havrilesky LJ. Promoting Same-Day Discharge for Gynecologic Oncology Patients in Minimally Invasive Hysterectomy. J Minim Invasive Gynecol. 2017 Sep-Oct;24(6):932-939. doi: 10.1016/j.jmig.2017.05.005. Epub 2017 May 10. PMID 28501452
- [Background] Kenton K, Pham T, Mueller E, Brubaker L. Patient preparedness: an important predictor of surgical outcome. Am J Obstet Gynecol. 2007 Dec;197(6):654.e1-6. doi: 10.1016/j.ajog.2007.08.059. PMID 18060968
- [Background] Brubaker L, Litman HJ, Rickey L, Dyer KY, Markland AD, Sirls L, Norton P, Casiano E, Paraiso MF, Ghetti C, Rahn DD, Kusek JW. Surgical preparation: are patients "ready" for stress urinary incontinence surgery? Int Urogynecol J. 2014 Jan;25(1):41-6. doi: 10.1007/s00192-013-2184-x. Epub 2013 Aug 3. PMID 23912506